CLINICAL TRIAL: NCT01412047
Title: A Post Marketing, Multi-Center, Trial to Measure Human Anti-Human Antibodies (HAHA) to Soliris (Eculizumab) in Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Paroxysmal Nocturnal Hemoglobinuria Human Anti-Human Antibodies Study
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: M07-003
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria; PNH
Keywords: Paroxysmal Nocturnal Hemoglobinuria; PNH; Human Anti-Human Antibody; HAHA; Soliris; eculizumab
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
How does long term treatment with Soliris affect HAHA in PNH patients?

DETAILED DESCRIPTION:
To determine the long term effect of Soliris (eculizumab) treatment on the presence of human anti-human antibodies (HAHA) in Paroxysmal Nocturnal Hemoglobinuria (PNH) patients.

ELIGIBILITY:
Inclusion Criteria:

* PNH patients who previously participated in study E05-001;
* Patients who have an eculizumab naive serum sample for comparison;
* Patients who currently used commerical Soliris;
* Patients who are willing and able to gie written informed consent.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with PNH previously enrolled in study E05-001, who have a eculizumab naive serum sample available for comparison, and who are currently receiving treatment with commerical Soliris.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
To summarize the proportion of patients with neutralizing HAHA antibodies. | Six (6) months

SECONDARY OUTCOMES:
To summarize the proportion of patients with non-neutralizing HAHA antibodies. | Six (6) months
To summarize the proportion of patients with increased hemolysis in setting of neutralizing HAHA antibodies. | Six (6) months

CONTACTS AND LOCATIONS:
Overall Officials: Camille Bedrosian, MD, Study Director — Alexion Pharmaceuticals, Inc.
Locations (14):
- United States (3):
  - University Park Hematology Oncology, Englewood, Colorado
  - Cleveland Clinic Florida, Weston, Florida
  - Maine Cancer Center of Medicine, Scarborough, Maine
- Melbourne, Australia
- Brussels, Belgium
- Paris, France
- Germany (2):
  - Universitatsklinikum Essen, Essen
  - Institut fur Klinische Transfusionmedizin und Immungenetick, Ulm
- Dublin, Ireland
- Italy (2):
  - Azienda Ospediliera Universitatia Careggi, Florence
  - Universita degli Studi di Napoli, Napoli
- Nijmegen, Netherlands
- Basel, Switzerland
- London, United Kingdom

IPD SHARING:
Plan to Share IPD: No